CLINICAL TRIAL: NCT01943526
Title: Ireland Natalizumab (TYSABRI®) Observational Program (iTOP)
Brief Title: Ireland Natalizumab (TYSABRI) Observational Program
Acronym: iTOP
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: TYS-IRL-11-4
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Ireland; Natalizumab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: natalizumab — Natalizumab will not be provided as a part of this study. Participants will receive natalizumab as prescribed by their treating physician.
  Other Names: Tysabri; BG00002

SUMMARY:
The objectives of this study are to assess the long-term safety and impact on disease activity and progression of natalizumab (Tysabri) in participants with relapsing remitting multiple sclerosis (RRMS) in a clinical practice setting.

DETAILED DESCRIPTION:
iTOP is a retrospective and prospective Irish observational study of participants receiving natalizumab, with each participant to be followed for 3 years. This study is designed to address the long-term safety profile and the long-term impact on disease activity and progression of natalizumab with marketed use. Collection of efficacy and safety data at 6- monthly intervals to coincide with regular clinic visits and routine clinical practice will therefore be undertaken during the iTOP observational period.

ELIGIBILITY:
Key Inclusion Criteria:

* Must give written informed consent and assent, as applicable.
* Decision to treat with natalizumab must precede enrollment.
* Patient characteristics and contraindications to treatment with natalizumab in accordance with prescribing information.
* Must be receiving natalizumab (Tysabri) for the treatment of RRMS in accordance with the natalizumab indication statement.
* Must have a documented diagnosis of Relapsing Remitting Multiple Sclerosis (RRMS).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RRMS who are being treated with natalizumab and patients who meet the criteria defined in the indication statement for prescription in Ireland. Existing patients will be enrolled retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing Serious Adverse Events (SAEs) | up to 3 years

SECONDARY OUTCOMES:
Disability progression as determined by Expanded Disability Status Scale (EDSS) | Up to 3 years
  Disability progression is defined as at least a 1.0 point increase on the EDSS from Baseline that is sustained over 6 months. The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
MS disease activity as determined by annualized relapse rate (ARR) | Up to 3 years
  A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement. New or recurrent neurological symptoms that occur less than 30 days following the onset of a protocol-defined relapse should be considered part of the same relapse.
MS disease activity as determined by distribution of the total number of relapses during the study | Up to 3 years
MS disease activity as determined by time to first relapse | Up to 3 years
MS disease activity as determined by number of participants with relapse | Up to 3 years
MS disability progression and MS disease activity summarized for subpopulations according to baseline characteristics | Up to 3 years
  Prognostic factors for disability progression and MS disease activity will be assessed in different participant cohorts stratified according to their baseline characteristics: Participant demographics including age, gender; Disease History, including diagnosis and duration at baseline; Baseline EDSS; Number of relapses within 1 and 2 years before baseline; MRI parameters at baseline; Prior use of disease modifying therapy, anti-neoplastic, immunosuppressant or immunomodulator therapy
MS disease activity as determined by MRI parameters | Up to 3 years
Evaluation of short-term disease outcomes as assessed by EDSS progression | Up to 1 year
Evaluation of short-term disease outcomes as assessed by occurrence of relapses | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- Ireland (5):
  - Research site, Cork, County Cork
  - Research site, Dublin, County Dublin
  - Research site, Galway, County Galway
  - Research site, Tralee, County Kerry
  - Research site, Sligo, County Sligo